CLINICAL TRIAL: NCT07243808
Title: Comparison of Mixed Reality and Ultrasound Localization Techniques for Surgical Stabilization of Rib Fractures
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202508142DINC
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Surgical Stabilization of Rib Fracture
Keywords: Ultrasound-guided localization; Mixed reality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mixed reality and Ultrasound Guided Localization: This cohort includes participants undergoing surgical stabilization of rib fractures (SSRF) who, as part of routine preoperative planning, receive both mixed reality (MR) and ultrasound surface marking before surgery. Investigators do not assign exposure; both methods are performed within the same participant to enable a within-subject comparison of localization accuracy (cm). Outcomes are abstracted from the medical record and outpatient clinic follow-up through about 90 days after surgery (e.g., localization accuracy by method, localization time, operative time, incision length, complications, pain scores, length of stay, wound healing).

SUMMARY:
The goal of this observational study is to compare two localization methods used before surgical stabilization of rib fractures (SSRF): mixed reality (MR) and ultrasound-guided.

Main Research Question Before SSRF, does MR help surgeons mark rib fracture locations more accurately (in centimeters) and faster than ultrasound-guided?

Participants After the study ends, all participants will keep follow-up at the thoracic surgery clinic. The team will record wound healing and pain scores for use in the observational study.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 80 years
2. Computed tomography (CT) demonstrates ≥3 rib fractures, and the patient meets indications for surgical stabilization of rib fractures (SSRF).
3. Able to understand the study and provide written informed consent.

Exclusion Criteria:

1. Uncorrected coagulopathy.
2. Known osteoporosis or pathologic fractures.
3. Respiratory failure or hemodynamic instability requiring emergent surgery.
4. Declines to participate or withdraws consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adults 18-80 years with CT-confirmed ≥3 rib fractures who meet indications for surgical stabilization of rib fractures (SSRF) at participating thoracic surgery services. Participants are managed under routine care and, as part of preoperative planning, receive both mixed reality (MR) and ultrasound surface marking to enable within-subject accuracy comparisons. Enrollment is prospective (non-probability sampling). Key exclusions include uncorrected coagulopathy, known osteoporosis or pathologic fractures, and respiratory failure or hemodynamic instability requiring emergent surgery.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-10-29 (Estimated)

PRIMARY OUTCOMES:
Rib fracture localization accuracy (cm) | Intraoperative assessment during the index SSRF procedure (immediately after fracture exposure and before plate fixation).
  Definition: For each participant and each method (mixed reality [MR; OpVerse] and ultrasound), accuracy is the absolute linear distance (cm) between the preoperative skin mark and the intraoperatively identified center of the fracture after exposure.
  Measurement: After skin incision and minimal soft-tissue dissection to expose the fracture line, the surgeon measures the shortest distance from the skin mark to the fracture center with a sterile ruler, recorded to 0.1 cm.
  Analysis note: Accuracy will be summarized per method, and a within-subject difference (MR minus ultrasound) will be calculated.
  Procedural note: If exposure is inadequate, the incision may be extended at the surgeon's discretion to safely perform SSRF; this does not change the measurement definition.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun DW, Zhai HX, Zhi JH, Chen KQ, Pang X, Xu M. Comparative efficacy of tunnel minimally invasive technique versus traditional open reduction and internal fixation for rib fractures. Eur J Med Res. 2025 Jul 9;30(1):603. doi: 10.1186/s40001-025-02864-1. PMID 40635080
- [Background] Zheng YA, Lee YC, Huang JY, Hsieh HY, Chen YS, Chiang XH, Han PH, Lin MW, Hsu HH, Hung YP, Chen JS. Enhancing three-dimensional anatomical understanding in complex thoracic surgery: a comparative study of OpVerse and Synapse 3D. Eur J Cardiothorac Surg. 2025 Mar 28;67(4):ezaf069. doi: 10.1093/ejcts/ezaf069. PMID 40163682
- [Background] Jung H, Raythatha J, Moghadam A, Jin G, Mao J, Hsu J, Kim J. RibMR - A Mixed Reality Visualization System for Rib Fracture Localization in Surgical Stabilization of Rib Fractures: Phantom, Preclinical, and Clinical Studies. J Imaging Inform Med. 2025 Oct;38(5):3279-3293. doi: 10.1007/s10278-024-01332-2. Epub 2024 Dec 20. PMID 39707113
- [Background] Magalhaes R, Oliveira A, Terroso D, Vilaca A, Veloso R, Marques A, Pereira J, Coelho L. Mixed Reality in the Operating Room: A Systematic Review. J Med Syst. 2024 Aug 15;48(1):76. doi: 10.1007/s10916-024-02095-7. PMID 39145896
- [Background] Lo HL, Lee JY, Lu CK, Lo OY, Lu CC, Tsai DL, Lin SY. Ultra minimally invasive surgical stabilization of Rib fractures (uMI-SSRF): reduction and fixation techniques to minimize the surgical wound. World J Emerg Surg. 2024 Nov 15;19(1):35. doi: 10.1186/s13017-024-00566-3. PMID 39548542
- [Background] Schots JP, Vissers YL, Hulsewe KW, Meesters B, Hustinx PA, Pijnenburg A, Siebenga J, de Loos ER. Addition of Video-Assisted Thoracoscopic Surgery to the Treatment of Flail Chest. Ann Thorac Surg. 2017 Mar;103(3):940-944. doi: 10.1016/j.athoracsur.2016.09.036. Epub 2016 Dec 7. PMID 27939010
- [Background] Martin TJ, Cao J, Benoit E, Kheirbek T. Optimizing surgical stabilization of rib fractures using intraoperative ultrasound localization. J Trauma Acute Care Surg. 2021 Aug 1;91(2):369-374. doi: 10.1097/TA.0000000000003262. PMID 33938512
- [Background] Fokin AA, Hus N, Wycech J, Rodriguez E, Puente I. Surgical Stabilization of Rib Fractures: Indications, Techniques, and Pitfalls. JBJS Essent Surg Tech. 2020 May 7;10(2):e0032. doi: 10.2106/JBJS.ST.19.00032. eCollection 2020 Apr-Jun. PMID 32944413
- [Background] Sermonesi G, Bertelli R, Pieracci FM, Balogh ZJ, Coimbra R, Galante JM, Hecker A, Weber D, Bauman ZM, Kartiko S, Patel B, Whitbeck SS, White TW, Harrell KN, Perrina D, Rampini A, Tian B, Amico F, Beka SG, Bonavina L, Ceresoli M, Cobianchi L, Coccolini F, Cui Y, Dal Mas F, De Simone B, Di Carlo I, Di Saverio S, Dogjani A, Fette A, Fraga GP, Gomes CA, Khan JS, Kirkpatrick AW, Kruger VF, Leppaniemi A, Litvin A, Mingoli A, Navarro DC, Passera E, Pisano M, Podda M, Russo E, Sakakushev B, Santonastaso D, Sartelli M, Shelat VG, Tan E, Wani I, Abu-Zidan FM, Biffl WL, Civil I, Latifi R, Marzi I, Picetti E, Pikoulis M, Agnoletti V, Bravi F, Vallicelli C, Ansaloni L, Moore EE, Catena F. Surgical stabilization of rib fractures (SSRF): the WSES and CWIS position paper. World J Emerg Surg. 2024 Oct 18;19(1):33. doi: 10.1186/s13017-024-00559-2. PMID 39425134
- [Background] Dehghan N, Nauth A, Schemitsch E, Vicente M, Jenkinson R, Kreder H, McKee M; Canadian Orthopaedic Trauma Society and the Unstable Chest Wall RCT Study Investigators. Operative vs Nonoperative Treatment of Acute Unstable Chest Wall Injuries: A Randomized Clinical Trial. JAMA Surg. 2022 Nov 1;157(11):983-990. doi: 10.1001/jamasurg.2022.4299. PMID 36129720
- [Background] Lian KH, Yang CC, Hu FC, Lin WY, Hsiao WL, Lin TH, Hu RH, Chen JS, Liao HC. Quality of life outcomes after surgical intervention in patients with multiple rib fractures: A prospective cohort study. Surgery. 2023 Apr;173(4):1066-1071. doi: 10.1016/j.surg.2022.12.006. Epub 2023 Jan 17. PMID 36658082
- [Background] Liu HY, Lin TH, Chen KC, Hsiao WL, Hu RH, Liao HC. Comparison between non-surgical and surgical management of rib fractures in major trauma patients without brain injuries. Am J Surg. 2023 Sep;226(3):350-355. doi: 10.1016/j.amjsurg.2023.05.025. Epub 2023 May 25. PMID 37263888
- [Background] Kao CC, Chen KC, Chiang XH, Chuang JH, Lu CW, Hsiao WL, Lin TH, Liao HC. Clinical outcomes of rib fracture stabilization and conservative treatment in a high-volume Asian trauma center: a propensity score-matched retrospective study. World J Emerg Surg. 2025 May 19;20(1):40. doi: 10.1186/s13017-025-00620-8. PMID 40390007
- [Background] Pieracci FM, Leasia K, Bauman Z, Eriksson EA, Lottenberg L, Majercik S, Powell L, Sarani B, Semon G, Thomas B, Zhao F, Dyke C, Doben AR. A multicenter, prospective, controlled clinical trial of surgical stabilization of rib fractures in patients with severe, nonflail fracture patterns (Chest Wall Injury Society NONFLAIL). J Trauma Acute Care Surg. 2020 Feb;88(2):249-257. doi: 10.1097/TA.0000000000002559. PMID 31804414